CLINICAL TRIAL: NCT00656487
Title: Translational Center on the Clinical Neurobiology of Cannabis Addiction
Brief Title: Clinical and Neurobiological Effects of Cannabis Dependence in Young Adults
Acronym: SCCAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DA024194; P20DA024194 (NIH)
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Cannabis Dependence; Cannabis Withdrawal
Keywords: Cannabis Dependence; Marijuana Dependence; Cannabis Withdrawal; Rimonabant; cannabinoid receptor type 1 (CB1) inverse agonist; Neuropsychology; functional magnetic resonance imaging (fMRI); Endocannabinoids; Cortisol
MeSH Terms: conditions — Marijuana Abuse | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cannabis-dependent rimonabant (Experimental): Cannabis dependent young adults administered rimonabant 90 mg at Day 0 and followed for 28 days post.
  Interventions: Drug: rimonabant
- Cannabis-dependent placebo (Placebo Comparator): Cannabis dependent young adults administered matched placebo at Day 0 and followed for 28 days post.
  Interventions: Drug: placebo
- Non-cannabis using control (No Intervention): Non-cannabis using demographically similar young adults followed for 28 days.

INTERVENTIONS:
Drug: rimonabant — double blind, placebo controlled, single 90 mg dose
  Other Names: CB1 receptor antagonist
  Arms: Cannabis-dependent rimonabant
Drug: placebo — matched placebo
  Arms: Cannabis-dependent placebo

SUMMARY:
The purpose of this study is to find out more about cognitive functioning in people who are cannabis dependent, relative to people who do not use cannabis, and how their brains process information after one month of not using cannabis. An additional goal is to characterize the severity of cannabis dependence using precipitated and naturalistic withdrawal with a double blind, placebo controlled, single administration of rimonabant. Research assessments occur bi-weekly throughout this 28 day study.

ELIGIBILITY:
Cannabis Dependent Subjects:

Inclusion Criteria:

* males or females 21-30 years of age
* meets Diagnostic and Statistical Manual (DSM-IV) diagnosis of Cannabis Dependence
* willing to be abstinent for 28 days during study
* smokes < 10 cigarettes per day
* drinks < 1 (female) or < 2 (male) per day

Exclusion Criteria:

* active suicide ideation
* meets DSM-IV diagnosis for dependence on other substances other than cannabis
* significant medical disorders
* pregnant women
* meets DSM-IV diagnosis for a major Axis I disorder other than cannabis dependence
* currently taking psychoactive medication

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2008-04-30 (Actual); Primary Completion 2010-12-28 (Actual); Study Completion 2011-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rimonabant: Participants were cannabis dependent and received a single 90 mg dose of rimonabant at baseline visit.
- Placebo: Participants were cannabis dependent and received matched placebo.
- Control: Participants were non-cannabis using controls.
Period: Overall Study
Arm/Group | Rimonabant | Placebo | Control
Started | 23 | 23 | 20
Completed | 21 | 19 | 20
Not Completed | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Per study design specifying that non-completers would be replaced to yield n=60 completers, two enrolled participants in the rimonabant group and four enrolled participants in the placebo group were not included in baseline (or additional) analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimonabant | Placebo | Control | Total
Number analyzed (Participants) | 21 | 19 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.33 (1.53) | 23.53 (2.76) | 24.15 (2.83) | 23.32 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 19
  Male | 15 | 12 | 14 | 41

OUTCOME MEASURES:

1. Primary Outcome: Withdrawal Symptom Severity on the Marijuana Withdrawal Checklist (MWC) at 28 Days Following Single Dose Administration of Rimonabant or Placebo, or Commencement of Monitoring, During the Double-Blind Period
Description: The MWC is a 28-item instrument that is used to assess the severity of frequently reported cannabis withdrawal symptoms. Each item on the measure is recorded as a severity rating between 0-3 where a zero indicates not present and a three indicates severe. The severity rating of each item was summed to obtain a single marijuana withdrawal severity score ranging between 0- 84. A lower score indicates less severe withdrawal.
Time Frame: Day 28
Population: One participant in the control group who completed monitoring during the double-blind portion of the trial did not complete a Marijuana Withdrawal Checklist at Day 28.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo | Control
Number analyzed (Participants) | 21 | 19 | 19
units on a scale | 6.62 (5.59) | 6.68 (7.87) | 1.05 (2.39)

2. Primary Outcome: Plasma Norepinephrine
Description: Blood samples were obtained and plasma concentrations were determined using validated enzyme-linked immunosorbent assay (ELISA) techniques at 28 days following single dose administration of rimonabant or placebo, or commencement of monitoring, during the double-blind period.
Time Frame: Day 28
Population: Five control participants who completed the double blind / monitoring portion of the trial did not have samples available for analysis at Day 28. Two participants did not have blood drawn; two additional participant sample results were not returned by the laboratory; and one participant did not return a result due to an ELISA kit error.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rimonabant | Placebo | Control
Number analyzed (Participants) | 21 | 19 | 15
ng/mL | 2.12 (1.14) | 2.04 (1.05) | 1.75 (0.84)

3. Primary Outcome: Plasma Cortisol
Description: as for outcome 2
Time Frame: Day 28
Population: Two control participants and one placebo participant who completed the double blind / monitoring portion of the trial did not have samples available for analysis at Day 28. The control participants did not have blood drawn; the placebo participant returned a non-detectable value.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Rimonabant | Placebo | Control
Number analyzed (Participants) | 21 | 18 | 18
ug/dL | 27.36 (15.03) | 19.29 (7.42) | 22.72 (15.21)

4. Primary Outcome: Change From Day 0 in Performance on the Cambridge Neuropsychological Test Automated Batteries Spatial Working Memory (CANTAB SWM) Strategy Score at Day 28
Description: The CANTAB SWM task is a validated computer-based testing instrument assessing the memory component of executive function. Strategy Score is an estimate of use of the most efficient strategy to complete the task. Scores range from 8-56; higher scores equate to poor use of the most efficient strategy. Change = (Day 28 Score - Day 0 Score). A more negative result indicates greater improvement.
Time Frame: Day 0 and Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo | Control
Number analyzed (Participants) | 21 | 19 | 20
units on a scale | -2.67 (4.15) | -1.37 (5.16) | -1.50 (3.62)

5. Primary Outcome: Change From Day 0 in Performance on the Cambridge Neuropsychological Test Automated Batteries Spatial Working Memory (CANTAB SWM) Total Errors at Day 28
Description: The CANTAB SWM task is a validated computer-based testing instrument assessing the memory component of executive function. Total Errors are a measure of performance and are unbounded. Change = (Day 28 Score - Day 0 Score). A more negative result indicates greater improvement.
Time Frame: Day 0 and Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo | Control
Number analyzed (Participants) | 21 | 19 | 20
units on a scale | -10.62 (13.46) | -1.95 (11.43) | -2.85 (9.36)

6. Primary Outcome: Change From Day 0 in Performance on the Cambridge Neuropsychological Test Automated Batteries Spatial Working Memory (CANTAB SWM) Mean Time To First Response at Day 28
Description: The CANTAB SWM task is a validated computer-based testing instrument assessing the memory component of executive function. Mean Time To First Response is a measure of latency and is unbounded. Change = (Day 28 Time - Day 0 Time). A more negative result indicates greater improvement.
Time Frame: Day 0 and Day 28
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Rimonabant | Placebo | Control
Number analyzed (Participants) | 21 | 19 | 20
milliseconds | -139.80 (414.68) | 420.24 (2262.39) | 22.01 (1438.16)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all ten study visits, an average duration of 28 days.
Description: Adverse events, both serious and other, were documented at all ten study visits by the Medical Assistant on the adverse experiences case report form.
Arm/Group | Rimonabant | Placebo | Control
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 10/23 | 10/23 | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rimonabant (N=23) | Placebo (N=23) | Control (N=20)
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Headache (Nervous system disorders) | 5 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No